CLINICAL TRIAL: NCT04471519
Title: An Adaptive Phase 1, Followed by Phase 2 Randomized, Double-blind, Multicenter Study to Evaluate the Safety, Reactogenicity, Tolerability, and Immunogenicity of BBV152 in Healthy Volunteers
Brief Title: Whole-Virion Inactivated SARS-CoV-2 Vaccine (BBV152) for COVID-19 in Healthy Volunteers
Acronym: BBV152
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bharat Biotech International Limited (Industry)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BBIL/BBV152-A/2020; Protocol No:BBIL/BBV152-A/2020 (Other: Bharat Biotech International Ltd)
Record Dates: First submitted 2020-07-11; First posted 2020-07-15 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: BBV152; COVID-19 vaccine; inactivated vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- BBV152A - Phase I (Experimental): 0.5 mL of Whole Virion Inactivated SARS-CoV-2 Vaccine [BBV152A], is a liquid vaccine administered intramuscularly twice at Day 0 and Day 14
  Interventions: Biological: BBV152A - Phase I
- BBV152B - Phase I (Experimental): 0.5 mL of Whole Virion Inactivated SARS-CoV-2 Vaccine [BBV152B], is a liquid vaccine administered intramuscularly twice at Day 0 and Day 14
  Interventions: Biological: BBV152B - Phase I
- BBV152C - Phase I (Experimental): 0.5 mL of Whole Virion Inactivated SARS-CoV-2 Vaccine [BBV152C], is a liquid vaccine administered intramuscularly twice at Day 0 and Day 14
  Interventions: Biological: BBV152C - Phase I
- Placebo - Phase I (Active Comparator): 0.5 mL of Placebo will be administered intramuscularly twice at Day 0 and Day 14.
  Interventions: Biological: Placebo - Phase I
- BBV152A - Phase II (Experimental): 0.5 mL of Whole Virion Inactivated SARS-CoV-2 Vaccine [BBV152A], is a liquid vaccine administered intramuscularly twice at Day 0 and Day 28.
  Interventions: Biological: BBV152A - Phase II
- BBV152B - Phase II (Experimental): 0.5 mL of Whole Virion Inactivated SARS-CoV-2 Vaccine [BBV152B], is a liquid vaccine administered intramuscularly twice at Day 0 and Day 28
  Interventions: Biological: BBV152B - Phase II

INTERVENTIONS:
Biological: BBV152A - Phase I — 0.5 ml of the vaccine will be administered intramuscularly twice at Day 0 and Day 14
  Arms: BBV152A - Phase I
Biological: BBV152B - Phase I — 0.5 ml of the vaccine will be administered intramuscularly twice at Day 0 and Day 14
  Arms: BBV152B - Phase I
Biological: BBV152C - Phase I — 0.5 ml of the vaccine will be administered intramuscularly twice at Day 0 and Day 14
  Arms: BBV152C - Phase I
Biological: Placebo - Phase I — 0.5 ml of the Placebo will be administered intramuscularly twice at Day 0 and Day 14
  Arms: Placebo - Phase I
Biological: BBV152A - Phase II — 0.5 ml of the vaccine will be administered intramuscularly twice at Day 0 and Day 28
  Arms: BBV152A - Phase II
Biological: BBV152B - Phase II — 0.5 ml of the vaccine will be administered intramuscularly twice at Day 0 and Day 28
  Arms: BBV152B - Phase II

SUMMARY:
Double blind, Multi-Centre study to evaluate the safety, reactogenicity, tolerability, and immunogenicity of three investigational vaccine groups and one placebo group in healthy volunteers who receive two intramuscular doses of BBV152 vaccine formulations and placebo. A total sample size of 755 healthy volunteers, with 375 and 380 volunteers in phase 1 and 2 studies, respectively.

A protocol amendment was made to evaluate a boosting regimen at the 6-month interval in the Phase 2 trial. At 6 months post-dose 2, participants who received the 6ug Algel-IMDG allocation were randomized equally to receive a third dose of BBV152 (6ug Algel-IMDG) or placebo.

DETAILED DESCRIPTION:
Phase 1 study

The study is designed to evaluate the safety, reactogenicity, tolerability, and immunogenicity of Four arms of healthy volunteers who receive two intramuscular doses of BBV152 vaccine formulations or Placebo. A total no of 375 subjects will be enrolled in 4:1 ratio.

This study will be conducted in a dose escalatory manner with a two-dose regimen fourteen days apart.

Phase 2 study

The study is designed to evaluate the safety, reactogenicity, tolerability, and immunogenicity of two arms of healthy volunteers who will receive two intramuscular doses of BBV152 vaccine formulations (BBV152-A & BBV152-B) in a 1:1 ratio with dosage schedule on Day 0 and Day 28.

A protocol amendment was made to evaluate a boosting regimen at the 6-month interval in the Phase 2 trial. At 6 months post-dose 2, participants who received the 6ug Algel-IMDG allocation were randomized equally to receive a third dose of BBV152 (6ug Algel-IMDG) or placebo. The investigator, participant and Sponsor were blinded to the allocation.

ELIGIBILITY:
Phase 1:

Inclusion Criteria

1. Ability to provide written informed consent.
2. Participants of either gender of age between ≥18 to ≤55 years.
3. Good general health as determined by the discretion of investigator (vital signs (heart rate ≥60 to≤100 bpm; blood pressure systolic ≥90 mm Hg and <140 mm Hg; diastolic ≥ 60 mm Hg and <90 mm Hg; oral temperature <100.4ºF), medical history, and physical examination).
4. Expressed interest and availability to fulfill the study requirements.
5. For a female participant of child-bearing potential, planning to avoid becoming pregnant (use of an effective method of contraception or abstinence) from the time of study enrolment until at least four weeks after the last vaccination
6. Male subjects of reproductive potential: Use of condoms to ensure effective contraception with the female partner from first vaccination until 3 months after last vaccination
7. Male subjects agree to refrain from sperm donation from the time of first vaccination until 3 months after last vaccination
8. Participants must refrain from blood or plasma donation from the time of first vaccination until 3 months after last vaccination
9. Agrees not to participate in another clinical trial at any time during the study period.
10. Agrees to remain in the study area for the entire duration of the study.
11. Willing to allow storage and future use of biological samples for future research.

Exclusion Criteria

1. History of any other COVID-19 investigational vaccination.
2. Unacceptable laboratory abnormality from screening (prior to first vaccination) or safety testing, as listed below [Abnormal Complete Blood Count (CBC), Random blood sugar level, Renal function test (serum urea and Creatinine), liver function tests, urine analysis report, Positive serology for hepatitis C or HIV antibody or hepatitis B surface antigen].

   (Subjects will be informed if their results are positive for hepatitis C, HIV 1 & 2 antibody or hepatitis B surface antigen (HBsAg) and will be referred to a primary care provider for follow up of these abnormal laboratory tests.)
3. Confirmed SARS-CoV-2 at the time of screening using RT-PCR and ELISA method.
4. Health care workers.
5. For women, a positive serum pregnancy test (during screening within 45 days of enrolment) or positive urine pregnancy test (within 24 hours of administering each dose of vaccine).
6. Temperature >38.0°C (100.4°F) or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis within three days prior to each dose of vaccine.
7. Medical problems as a result of alcohol or illicit drug use during the past 12 months.
8. Receipt of an experimental agent (vaccine, drug, device, etc.) within 60 days before enrollment or expects to receive an investigational agent during the study period.
9. Receipt of any licensed vaccine within four weeks before enrolment in this study.
10. Known sensitivity to any ingredient of the study vaccines, or a more severe allergic reaction and history of allergies in the past.
11. Receipt of immunoglobulin or other blood products within the three months prior to vaccination in this study.
12. Immunosuppression as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
13. Long-term use (> 2 weeks) of oral or parenteral steroids (glucocorticoids) or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding six months (nasal and topical steroids are allowed).
14. Any history of hereditary angioedema or idiopathic angioedema.
15. Any history of anaphylaxis in relation to vaccination.
16. Any history of albumin-intolerance.
17. Pregnancy, lactation, or willingness/intention to become pregnant during the study.
18. History of any cancer.
19. History of psychiatric severe conditions likely to affect participation in the study.
20. A bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder, or prior history of significant bleeding or bruising following IM injections or venepuncture.
21. Any other serious chronic illness requiring hospital specialist supervision.
22. Chronic respiratory diseases like severe acute respiratory syndrome (SARS), including mild asthma.
23. Chronic cardiovascular disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, and neurological illness
24. Morbidly obese (BMI≥35 kg/m2) or underweight (BMI ≤18 kg/m2).
25. Living in the same household of any COVID-19 positive person.
26. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.

    Re-Vaccination Exclusion Criteria
27. Pregnancy.
28. Anaphylactic reaction following administration of the investigational vaccine.
29. Virologically confirmed cases of COVID-19

Phase 2:

Inclusion Criteria

1. Ability to provide written informed consent (Audio video consent for vulnerable subjects).
2. Participants of either gender of age between ≥12 to ≤ 65 years.
3. Good general health as determined by the discretion of investigator (vital signs (heart rate ≥60 to≤100 bpm; blood pressure systolic ≥90 mm Hg and <140 mm Hg; diastolic ≥ 60 mm Hg and <90 mm Hg; oral temperature <100.4ºF), medical history, and physical examination).
4. Expressed interest and availability to fulfill the study requirements.
5. For a female participant of child-bearing potential, avoid becoming pregnant (use of an effective method of contraception or abstinence) from the time of study enrolment until at least four weeks after the last vaccination and agrees not to participate in another clinical trial at any time during the study period.
6. Male subjects of reproductive potential: Use of condoms to ensure effective contraception with the female partner from first vaccination until 3 months after last vaccination
7. Male subjects agree to refrain from sperm donation from the time of first vaccination until 3 months after last vaccination
8. Participants must refrain from blood or plasma donation from the time of first vaccination until 3 months after last vaccination.
9. Agrees to remain in the study area for the entire duration of the study.
10. Willing to allow storage and future use of biological samples for future research.

Exclusion Criteria

1. History of any other COVID-19 investigational vaccination.
2. Confirmed SARS-CoV-2 at the time of screening using RT-PCR and ELISA method.
3. Health care workers.
4. Positive urine pregnancy test (within 24 hours of administering each dose of vaccine).
5. Temperature > 38.0°C (100.4°F) or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis within three days prior to each dose of vaccine.
6. Medical problems as a result of alcohol or illicit drug use during the past 12 months.
7. Receipt of an experimental agent (vaccine, drug, device, etc.) within 60 days before enrolment or expects to receive an investigational agent during the study period.
8. Receipt of any licensed vaccine within four weeks before enrolment in this study.
9. Known sensitivity to any ingredient of the study vaccines, or a more severe allergic reaction and history of allergies in the past.
10. Receipt of immunoglobulin or other blood products within the three months prior to vaccination in this study.
11. Immunosuppression as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
12. Long-term use (> 2 weeks) of oral or parenteral steroids (glucocorticoids) or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding six months (nasal and topical steroids are allowed).
13. Any history of hereditary angioedema or idiopathic angioedema.
14. Any history of anaphylaxis in relation to vaccination.
15. Any history of albumin-intolerance.
16. Pregnancy, lactation, or willingness/intention to become pregnant during the study.
17. History of any cancer.
18. History of psychiatric severe conditions likely to affect participation in the study.
19. A bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder, or prior history of significant bleeding or bruising following IM injections or venepuncture.
20. Any other serious chronic illness requiring hospital specialist supervision.
21. Chronic respiratory diseases like severe acute respiratory syndrome (SARS), including mild asthma.
22. Chronic cardiovascular disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, and neurological illness
23. Morbidly obese (BMI≥35 kg/m2) or underweight (BMI ≤18 kg/m2).
24. Living in the same household of any COVID-19 positive person.
25. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.

    Re-Vaccination Exclusion Criteria
26. Pregnancy.
27. Anaphylactic reaction following administration of the investigational vaccine.
28. Virologically confirmed cases of COVID-19.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 755 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Phase 1: Occurrence of adverse events and Serious Adverse events | Through study completion, an average of 6 months
  Safety
Phase 2: Evaluation of Neutralizing Antibody Titers | Through study completion, an average of 6 months
  Pre- and Post-vaccination immune response

SECONDARY OUTCOMES:
Phase 1: Evaluation of Neutralizing Antibody Titers | Through study completion, an average of 6 months
  Pre- and Post-vaccination immune response
Phase 2: Occurrence of adverse events and Serious Adverse events | Through study completion, an average of 6 months
  Safety
Phase 2: Evaluation of Neutralizing Antibody Titers | Through study completion, an average of 6 months
  Post-vaccination immune responses comparing two-dose and three dose regimens

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Savita Verma, MBBS, MD, Principal Investigator — PGIMS, Rohtak; Dr. Sanjay Kumar Rai, MBBS, MD, Principal Investigator — All India Institute of Medical Sciences, Delhi; Dr. Chandramani Singh, MBBS, MD, Principal Investigator — All India Institute of Medical Sciences; Dr. Ajeeth Pratap Singh, MBBS, MD, Principal Investigator — Rana Hospital and Trauma Centre, Gorakhpur; Dr. Satyajit Mohapatra, MBBS, MD, Principal Investigator — SRM Hospital and Research Centre, Chennai; Dr. Prabhakar Reddy, MBBS, MD, Principal Investigator — Nizams Institute of Medical Sciences, Hyderabad; Dr. Venkata Rao, MBBS, MD, Principal Investigator — IMS & SUM Hospital, Orissa; Dr. Jitendra Kushwaha, MBBS, MD, Principal Investigator — Prakhar Hospital, Kanpur; Dr. Sagar Vivek Redkar, MBBS, MD, Principal Investigator — Redkar Hospital and Research Center, Goa; Dr. Amit Bhate, MBBS, MD, Principal Investigator — Jeevan Rekha Hospital, Belguam; Dr. Chadrashekar Gillukar, MBBS, MD, Principal Investigator — Gillukar Multispeciality Hospital, Nagpur; Dr Vasudev R, MBBS, MD, Principal Investigator — King George Hospital
Locations (12):
- India (12):
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - All India Institute of Medical Sciences, Patna, Bihar
  - Pt BD SHARMA,PGIMS/UHS, Rohtak, Haryana
  - Jeevan Rekha Hospital, Belagavi, Karnataka
  - Gillukar Multispeciality Hospital, Nagpur, Maharashtra
  - All India Institute of Medical Sciences, Delhi, New Delhi
  - Institute of Medical Sciences and SUM Hospital, Bhubaneswar, Odisha
  - SRM Hospital & Research center, Chennai, Tamil Nadu
  - Nizam's Institute of Medical Sciences, Hyderabad, Telangana
  - Rana Hospital and Trauma Center, Gorakhpur, Uttar Pradesh
  - Prakhar Hospital, Kanpur, Uttar Pradesh
  - Redkar Hospital and Research Centre, Goa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vadrevu KM, Ganneru B, Reddy S, Jogdand H, Raju D, Sapkal G, Yadav P, Reddy P, Verma S, Singh C, Redkar SV, Gillurkar CS, Kushwaha JS, Mohapatra S, Bhate A, Rai SK, Ella R, Abraham P, Prasad S, Ella K. Persistence of immunity and impact of third dose of inactivated COVID-19 vaccine against emerging variants. Sci Rep. 2022 Jul 14;12(1):12038. doi: 10.1038/s41598-022-16097-3. PMID 35835822
- [Derived] Ella R, Reddy S, Jogdand H, Sarangi V, Ganneru B, Prasad S, Das D, Raju D, Praturi U, Sapkal G, Yadav P, Reddy P, Verma S, Singh C, Redkar SV, Gillurkar CS, Kushwaha JS, Mohapatra S, Bhate A, Rai S, Panda S, Abraham P, Gupta N, Ella K, Bhargava B, Vadrevu KM. Safety and immunogenicity of an inactivated SARS-CoV-2 vaccine, BBV152: interim results from a double-blind, randomised, multicentre, phase 2 trial, and 3-month follow-up of a double-blind, randomised phase 1 trial. Lancet Infect Dis. 2021 Jul;21(7):950-961. doi: 10.1016/S1473-3099(21)00070-0. Epub 2021 Mar 8. PMID 33705727
- [Derived] Yadav PD, Ella R, Kumar S, Patil DR, Mohandas S, Shete AM, Vadrevu KM, Bhati G, Sapkal G, Kaushal H, Patil S, Jain R, Deshpande G, Gupta N, Agarwal K, Gokhale M, Mathapati B, Metkari S, Mote C, Nyayanit D, Patil DY, Sai Prasad BS, Suryawanshi A, Kadam M, Kumar A, Daigude S, Gopale S, Majumdar T, Mali D, Sarkale P, Baradkar S, Gawande P, Joshi Y, Fulari S, Dighe H, Sharma S, Gunjikar R, Kumar A, Kalele K, Srinivas VK, Gangakhedkar RR, Ella KM, Abraham P, Panda S, Bhargava B. Immunogenicity and protective efficacy of inactivated SARS-CoV-2 vaccine candidate, BBV152 in rhesus macaques. Nat Commun. 2021 Mar 2;12(1):1386. doi: 10.1038/s41467-021-21639-w. PMID 33654090
- [Derived] Ella R, Vadrevu KM, Jogdand H, Prasad S, Reddy S, Sarangi V, Ganneru B, Sapkal G, Yadav P, Abraham P, Panda S, Gupta N, Reddy P, Verma S, Kumar Rai S, Singh C, Redkar SV, Gillurkar CS, Kushwaha JS, Mohapatra S, Rao V, Guleria R, Ella K, Bhargava B. Safety and immunogenicity of an inactivated SARS-CoV-2 vaccine, BBV152: a double-blind, randomised, phase 1 trial. Lancet Infect Dis. 2021 May;21(5):637-646. doi: 10.1016/S1473-3099(20)30942-7. Epub 2021 Jan 21. PMID 33485468